CLINICAL TRIAL: NCT00605332
Title: Crux Biomedical Evaluation of the Crux Inferior Vena Cava Filter System - ("Retrieve")
Brief Title: Crux Biomedical IVC Filter - Evaluation of the Crux Inferior Vena Cava Filter System (Retrieve)
Acronym: Retrieve
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Crux Biomedical (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: RETRIEVE I; G070035
Record Dates: First submitted 2008-01-02; First posted 2008-01-31 (Estimated); Last update posted 2012-08-06 (Estimated); Status verified 2012-08

CONDITIONS: Pulmonary Embolism
MeSH Terms: conditions — Pulmonary Embolism | interventions — Vena Cava Filters

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): Investigative Device (Crux Biomedical IVC Filter) will be evaluated for its ability to capture thrombus for the prevention of pulmonary embolism.
  Interventions: Device: inferior vena cava filter

INTERVENTIONS:
Device: inferior vena cava filter — Crux Biomedical IVC Filter
  Other Names: No other names

SUMMARY:
This is an open label, non-randomized, prospective, multicenter study.

ELIGIBILITY:
Inclusion Criteria:

Patients for this study must meet the following inclusion criteria to be eligible for enrollment:

1. The patient is >18 years of age.
2. Patient is considered a candidate for the IVCF under one of the following indications:

   * Proven PE
   * Recurrent PE despite adequate anticoagulation
   * Contraindication to anticoagulation
   * Inability to achieve/maintain therapeutic anticoagulation
   * Iliocaval DVT
   * Large, free-floating proximal (i.e. ileofemoral) DVT
   * Massive PE treated with thrombolysis/thrombectomy
   * Chronic PE treated with thrombectomy
   * Protection during thrombolysis for iliocaval DVT
   * PE with limited cardiopulmonary reserve
   * Poor compliance with anticoagulant medications
   * High risk of injury worsened by anticoagulation (e.g., ataxia, falls)
   * Multi-trauma patient with high risk of PE
   * Surgical patients at high risk of PE
   * Medical condition with high risk of PE
3. Patient has a vena cava diameter of 17-28mm.
4. The patient or legal guardian has been informed of the nature of the study and agrees to its provisions and has provided informed written consent.
5. The patient is willing to be available for the appropriate follow-up for the duration of the study.
6. The patient has suitable IVC anatomy that would allow infra-renal placement of the filter.

Exclusion Criteria:

Patients who have ANY of the following exclusion criteria are NOT eligible for the study:

1. The patient has one of the following conditions:

   * Renal vein thrombosis
   * IVC thrombosis extending to renal veins
   * Duplicate IVC
   * Gonadal vein thrombosis
   * Requires supra-renal filter placement
2. The patient has an uncontrolled infectious disease.
3. The patient is at risk for aseptic PE.
4. Patient has uncontrollable coagulopathy.
5. Patient has an existing IVCF.
6. The patient has a life expectancy of less than 6 months.
7. The patient is pregnant.
8. The patient has a condition that inhibits radiographic visualization of the IVC.
9. The patient has a known allergy or intolerance to polytetrafluoroethylene (PTFE) or Nitinol.
10. The patient has a known hypersensitivity to contrast which cannot be pre-treated.
11. The patient's access vessels preclude safe insertion of the delivery system.
12. The patient is participating in another device or drug study. Patient must have completed the follow- up phase of any previous study at least 30 days prior to enrollment into this trial. The patient may only be enrolled in this study once.
13. The patient is unable and/or unwilling to cooperate with study procedures or required follow-up visits.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2007-10; Primary Completion 2008-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Primary Efficacy Objective: To describe the clinical utility of the Crux IVCF by the following criteria: Absence of a recurrent PE and IVC thrombosis related to the Crux IVCF. | 30 days post implant, 30 days post retrieval. Patients with indwelling filters will return 1 and 6 months post implant procedure.

SECONDARY OUTCOMES:
Primary Safety Objective: To estimate the proportion of patients who experience device/procedure related complications associated with the Crux IVCF. | 30 days post implant procedure and 30 days post retrieval procedure. Patients with indwelling filters will return 1 and 6 months post implant procedure.

CONTACTS AND LOCATIONS:
Overall Officials: David Rosenthal, MD, Principal Investigator — Atlanta Vascular Specialists; Mel Schatz, Study Director — Crux Biomedical